CLINICAL TRIAL: NCT03277911
Title: Thyroid Dysfunction and Dyslipidemia in Patients With Chronic Kidney Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Elewa Ahmed, Resident of clinical pathology department, Assiut University
Other Study IDs: Clincal Pathology
Record Dates: First submitted 2017-09-05; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: CKD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Early diagnosis of thyroid and lipid disorders by regular screening, and treatment of such disorders in CKD patients may be highly beneficial to slow progression of CKD. The study will be conducted to investigate thyroid function and lipid profile in patients with chronic kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease[CKD] is becoming a serious health problem.The number of people with impaired renal function is rapidly rising, especially in industrialized countries. It is increasing rapidly worldwide at an annual growth rate of 8%. Chronic kidney disease [CKD] is defined as kidney disease that has been present for months to years. Chronic kidney disease [CKD] is a complex disease impacting more than twenty million individuals. Progression of CKD is associated with a number of serious complications, including increased incidence of cardiovascular disease, hyperlipidemia, anemia and metabolic bone disease .CKD patients should be assessed for the presence of these complications and receive optimal treatment to reduce their morbidity and mortality .

CKD affects thyroid function in many ways, including low thyroid circulating hormone levels, altered peripheral hormone metabolism, insufficient binding to carrier proteins, reduced tissue thyroid hormone content and altered iodine storage in the thyroid gland.Thus,inCKD,thyroid hormone metabolism is impaired. . Hypothyroidism in patients with renal failure causes many metabolic and clinical problems, and both these diseases can mutually exacerbate their disturbances.. Chronic kidney disease has been known to affect thyroid hormones metabolism .Low serum level of T3 and T4 are most remarkable laboratorial finding. A high incidence of goiter and nodules on thyroid ultrasonography has been reported in patients with end stage renal failure[ESRF]. CKD is often associated with dyslipidemia. Several factors contribute to these changes. Patient with CKD have a reduction in the activity of lipoprotein lipase and hepatic triglyceride lipase. This interferes with uptake of triglyceride rich Apo lipoprotein B containing lipoprotein by the liver and in peripheral tissue, yielding increased circulation of these atherogenic lipoproteins. Early diagnosis of thyroid and lipid disorders by regular screening, and treatment of such disorders in CKD patients may be highly beneficial to slow progression of CKD.

ELIGIBILITY:
Inclusion criteria:

1. Patients with CKD stage (1-5).
2. Not known thyroid disorders.
3. Not in lipid lowering agents.

Exclusion Criteria:

1. Patients with known thyroid disorders, on medication affecting thyroid function and lipid lowering agents are excluded from the study.
2. CKD patients who were or underwent previous dialysis.
3. Nephrotic syndrome.
4. Obesity.
5. Patients on estrogens, corticosteroids, antithyroid drugs, dietary supplements.
6. Pregnant woman

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will be conducted on 80 patients with chronic kidney disease at Assuit University hospital to investigate thyroid function and lipid profile in patients with CKD of stages (1-5) and 20 subjects as a normal control. A total of newly diagnosed and known CKD cases of stage 1-5 will be included in the study.
  Sample Size Calculation:
  * Group I: Controls-20 age and sex matched normal individuals.
  * Group II: Cases -40 patients with stage 1-3.
  * Group III: Cases -40 patients with stage 4 and 5
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-10 (Estimated); Primary Completion 2018-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
The study will be conducted to investigate thyroid function in patients with chronic kidney disease | one year
  serum urea, creatinine, , triiodothyronine [T3], free thyroxin [T4], thyroid stimulating hormones [TSH]
The study will be conducted to investigate lipid profile in patients with chronic kidney disease | one year
  serum urea, creatinine,high density lipoprotein [HDL] cholesterol, low density cholesterol, total cholesterol, triglyceride